CLINICAL TRIAL: NCT01239550
Title: Making an "Obese"Brain(and Body)Lean: Insulin Detemir,Monoamines,and Reward
Brief Title: Insulin Detemir in Obesity Management
Acronym: IDIOM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Kevin Niswender, Associate Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KDN2010
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Obesity
Keywords: Insulin; Detemir; Dopamine, brain,neurotransmitter; Diabetes; Obesity; Neurotransmitters
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Insulin Resistance | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Detemir Treatment (Experimental): Insulin detemir treatment: Insulin detemir will be administered subcutaneously, once daily. Dose ranges from approximately 0.1 U/kg up to 0.6 u/kg or higher. The dosing regimen will employ a strategy similar to the "303"algorithm, where, with close interaction with study personnel (rather than self-titration), bedtime insulin dosing will be titrated up by 3 units until AM fasting sugars within the prescribed protocol range are achieved (90-110 mg/dl). Subjects will have contact with study personnel on weekly basis for glycemia monitoring and adjustments. Similarly, documented hypoglycemia (blood sugars less than 70) will trigger a dose reduction, and it is expected that with weight loss, tolerable insulin dosages will drift downward. The treatment period is 24 weeks.
  Interventions: Drug: Detemir
- Comparator: No insulin (No Intervention): The main hypothesis is that "diabetes can be changed " with early and careful insulinization capturing effects on brain function ultimately leading to weight loss. . Seek to determine in a quantitative manner whether insulin detemir restores brain dopamine neurotransmission, a control group not treated with insulin is required. The strength of this study is our ability to test the specific molecular (D2R, DAT, functional MRI responses) and integrated output (functional brain responses, mood, cognitive function, reward responses etc.) of CNS dopaminergic pathways in order to shed unprecedented light upon mechanisms of detemir action in obesity and diabetes.

INTERVENTIONS:
Drug: Detemir — Subjects randomized to insulin detemir treatment group will receive the basal insulin in a 3 mL. Flex Pen® containing 300 units of insulin. insulin detemir once daily administered with the evening meal (dinner) or at bedtime as add-on to their oral antihyperglycemia (see inclusion/exclusion criteria) meds throughout the 24 week treatment period. The goal of insulin therapy is to achieve near normoglycemia with a low rate of hypoglycaemic episodes.
  Insulin injections will be given subcutaneously preferably in the thigh or abdomen.
  Other Names: Levemir
  Arms: Insulin Detemir Treatment

SUMMARY:
The purpose of this study is to evaluate the effects of the medication insulin detemir on weight, brain function and mood, and on blood vessel and other risk factors for heart disease. The study will compare how diet and insulin detemir affect areas of the brain that are involved in food intake and the sense of pleasure people get from eating.

Participants will be randomized into one of 2 groups. Group 1 will follow a low calorie diet only. Group 2 will follow a low calorie diet and take insulin detemir.

The study is 26 weeks in length and include outpatient visits, inpatient visits, phone and email contact, questionnaires, diary collection, blood draw and procedures involving MRI and PET scans. There are 4 inpatient visits at the Vanderbilt Clinical Research Center (CRC). The inpatient visits require a one night 2 day stay on the CRC at Weeks 2, 6, 16, 26. During the weekly and bi-weekly outpatient visits participants will meet with the study nurse and dietitian.

DETAILED DESCRIPTION:
Together with obesity, diabetes is epidemic in the US (20) and worldwide (21). Increased body weight is both a risk factor for diabetes (22) and a consequence of initiation and intensification of insulin therapy, as illustrated in landmark diabetes control trials (1-3). Weight gain can worsen insulin resistance leading to higher insulin requirements, and, thus perpetuates a vicious cycle (36), the ultimate effect of which may be to further enhance metabolic risk (15, 35). For example, an analysis of the diabetes control and complications trial (DCCT) revealed that the highest quartile of weight gain in the intensive treatment led to hyperlipidemia and increased blood pressure; i.e. metabolic syndrome (35). Thus, while glycemic control is clearly a critical metabolic target in diabetes outcomes, additional considerations, including body weight (adiposity) and weight gain, are of fundamental importance in the clinical management of a complex disease such as diabetes. Of course, overweight and obesity are clearly a critical risk factor for the development of type II diabetes in the first place (10), and further weight gain generates significant negative "biofeedback" to the patient and physician struggling to achieve control(33).

Mechanisms involved in weight gain on insulin therapy are incompletely understood: hypoglycemia is potent stimulus to feed (11), improving glycemic control reverses the negative energy balance associated with glycosuria (loss of energy as glucose through the urine), and insulin is clearly a potent anabolic hormone in peripheral tissues (37). In contrast to ample evidence associating insulin therapy with weight gain, a distinct body of evidence indicates that insulin functions as an adiposity negative feedback signal to the brain (23) and limits food intake and weight gain. It is now generally accepted that insulin plays an important role in the neural control of energy homeostasis (matching of caloric intake to energy expenditure to maintain body weight) as well as glucose homeostasis via such neural effects (23). Of course, as will be further discussed, insulin has numerous effects in the CNS ranging from modulation of reward (12), cognition (31), and mood (32). Indeed, the overarching hypothesis of this study is that insulin modulates brain function in a manner that is beneficial.

Food reward can loosely be described as the processes involved in liking, wanting, and learning to acquire food and each of these aspects represent separate but overlapping neuropsychological substrates. To put it even more simply, reward is the sense of satisfaction or pleasure derived from eating. Food reward has sensory, integrative, and motor components, all of which contribute to consummatory behaviors (38). Relevant to the focus of this particular study, is the monoamine neurotransmitter dopamine, which is heavily involved in the generation of food reward. Insulin, a signal generated in response to food intake, functions to decrease, or control food reward(12).

Reward, defined as the sense of satisfaction, or indeed, pleasure that results from feeding is an increasingly recognized and potentially potent influence over food intake that shares neuoranatomical and neurochemical correlates with substance abuse (although with clear differences as well). Although other neurotransmitters (in particular opioids and endocannabinoids) are involved in reward, the monoamine neurotransmitter, dopamine (DA) has been strongly implicated in mediating reward from food (and other stimuli). The midbrain is particularly rich in dopamine neurons, originating in the ventral tegmental area (VTA) that project to both ventral (nucleus accumbens, NAc) and dorsal (caudate and putamen) striatum, brain areas that integrate and subserve reward and food seeking behaviors. While the circuitry involved in feeding and reward is complex, these discreet brain areas (dorsal and ventral striatum) are heavily dopaminergic, implicated in reward, and are brain areas that our group has a great deal of expertise in studying.

Dopamine is secreted into the synapse from pre-synaptic nerve terminals and either binds to and activates dopamine receptor signaling, or is cleared from the synaptic cleft by a specific transporter molecule. The dopamine receptor of interest for this study is the D2 receptor, as it has been well studied and is the isoform involved in feeding. Similarly, the dopamine transporter has been well studied, plays a critical role in dopamine neurotransmission, and is regulated by insulin. In this study we will utilize PET radioligands to quantify expression of D2 receptors. We will additionally utilize functional brain imaging (functional magnetic resonance imaging (fMRI)) to quantify changes in dopamine circuits in response to food cues (visual images of obesogenic food) and in response to a probe of dopamine transporter function.

Although weight-gain on insulin initiation or intensification is common, numerous reports in randomized, controlled human clinical trials describe attenuation of this effect with the basal insulin analogue, detemir ((17), reviewed in (18)). Intriguingly, the observed weight sparing effects of detemir appear to be amplified in the most obese (18), i.e. the effects of detemir are evident and even amplified in a situation in which insulin resistance is most severe. This scenario is entirely consistent with our overarching hypotheses described throughout. The current study will utilize insulin detemir as a tool to understand weight effects of insulin mediated by CNS effects and to identify the mechanisms involved in the observed weight sparing effect.

Insulin detemir was approved by the FDA for the treatment of diabetes in 2005. Detemir is a long-acting, basal insulin analogue with unique pharmacological properties that we believe confers the capacity to regulate brain insulin sensitive processes. Compared to regular human insulin, detemir has one amino acid deleted, and a medium chain fatty acid conjugated to amino acid B29. Conjugation of this fatty acid confers prolonged absorption from the subcutaneous depot as it mediates polymerization and slow release. Additionally the fatty acid confers albumin binding in the plasma, further increasing the half-life, and providing a second buffering mechanism for prolongation of duration of action. We hypothesize that this fatty acid additionally confers enhanced transport into the CNS and/or, enhanced signaling through the insulin receptor in the context where insulin resistance is established. In the clinical development program, insulin detemir was noted to cause significantly less weight gain, and from a safety perspective is also associated with less hypoglycemia.

Rationale for this study. Firstly, dopamine neurotransmission underlies reward. Several high visibility studies in humans provide proof-of-principle data supporting the hypothesis that defects in dopamine homeostasis contribute to the pathophysiology of obesity (40, 41). By PET imaging, dopamine D2 receptor availability (radioligand binding potential) was reduced in a BMI dependent fashion; i.e. with increased body mass, less dopamine D2 receptor is available in the brain for dopamine signaling (leading to reduced dopamine signaling; hypodopaminergia). Similarly, brain activation, as measured by functional MR imaging (using techniques similar to those utilized herein), was reduced in obese individual who possess polymorphisms in genes regulating dopamine signaling. This work, together with an ever expanding body of preclinical work indicates that obesity is a chronic state of reduced dopamine signaling, or hypodopaminergia; indeed this condition has been termed "hypodopaminergic reward deficiency syndrome." As our preliminary data supports dopamine neurotransmission is under regulatory influence by insulin; insulin regulates intracellular trafficking of the transporter (analogous to insulin regulation of glucose transporter trafficking), and this trafficking is required to maintain the fidelity of dopamine signaling via the D2 receptor

ELIGIBILITY:
Inclusion criteria:

1. Informed consent obtained before any trial-related activities
2. Age at study entry is between 31-60 years of age
3. Body Mass index (BMI) between 30-49 kg/m2 using measured height and weight
4. Body weight <350lbs (MRI table limit)
5. Stable body weight during the previous 3 months with a less than 5 pounds self -reported weight change
6. Type 2 diabetes, insulin naïve (except for use during gestational diabetes) on either metformin, sitagliptin, or dipeptidyl-4 inhibitor (sitagliptin or saxagliptin), or a thiazolidines (rosiglitazone or pioglitazone)
7. HbA1c level between ~6-8%
8. Lives in a community dwelling and has a telephone
9. Agrees to avoid alcohol and exercise within 48 hours of CRC visits, and to comply with the dietary/stimulant restrictions for 48 hours before PET and fMRI studies.
10. Able and willing to follow prescribed menus plans

Exclusion Criteria:

1. Known or suspected hypersensitivity to study drug (insulin detemir)
2. Significant co-morbidities including cardiovascular disease, atherosclerotic disease, pulmonary disease, metabolic disease, liver or renal insufficiency
3. Significant pathologic finding on MRI (research MRI scans are not clinical scans and are not standardly read by a neuroradiologist, but if an overt anomaly is noted by study personnel, an advisory read will be obtained and the patient will be provided with the information for follow-up with his/her physician).
4. Clinically significant abnormalities on screening EKG
5. History of Substance Abuse, including but not exclusive to alcohol, cocaine, marijuana, heroin, nicotine
6. Any tobacco use in last 3 months
7. History of psychiatric disorder deemed too severe to permit participation (PI discretion) including subjects with a lifetime history of lifetime Psychotic Disorder (Schizophrenia, Schizoaffective, Psychosis NOS) or Bipolar Disorder, suicide attempt or history of any suicidal behavior or history within the past 6 months of Post Traumatic Stress Disorder, Generalized Anxiety Disorder
8. Long term use of steroids or medications that may cause weight gain within 3 months of study or in foreseeable need (e.g. uncontrolled asthma or rheumatologic disorder).
9. Inability to abstain from alcohol, physical exercise or > 1 cup of coffee or equivalent daily for 2 days prior to imaging studies
10. Any contraindication which would interfere with MRI or PET studies, e.g. claustrophobia, cochlear implant, metal fragments in eyes, cardiac pacemaker, neural stimulator, tattoos with iron pigment and metallic body inclusions or other metal implanted in the body
11. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (abstinence or the following methods: diaphragm with spermicide, condom with spermicide by male partner, intrauterine device, sponge, spermicide, Norplant, Depo-Provera or oral contraceptives)
12. History of uncontrolled thyroid disease evidenced by TSH outside normal range
13. Obesity induced by other endocrinologic disorders (e.g. Cushing Syndrome, Polycystic ovarian syndrome)
14. Previous surgery for weight loss
15. High level aerobic activity such as running for longer than 60 minutes more than 2 times a week regularly in last 3months
16. Significant eating disorder or dietary restraints as determined by three factor eating questionnaire (TFEQ)
17. Appetite reducing diet supplement or herbal supplement use in last 6 months
18. . Food allergy or diet restrictions that would interfere with balanced intake and caloric goals.
19. Dietary supplements of such as EPA, DHA or omega-3 fatty acids.
20. Daily intakes of coffee, black tea and other caffeinated beverages will be assessed and subjects who consume the equivalent of >4 cups coffee or black tea/day at baseline will be excluded
21. Any condition felt by PI or co-investigators to interfere with ability to complete the study

Ages: 31 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-04; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Low dose basal insulin detemir will potentiate weight loss in obese patients with type 2 diabetes mellitus undergoing a hypocaloric diet intervention by improving dopamine signaling | 26 weeks
  Determine if low dose basal insulin detemir potentiates loss of total body weight and adipose tissue in obese patients with type 2 diabetes mellitus undergoing a hypocaloric diet intervention

SECONDARY OUTCOMES:
Neuropsychiatric functions | 26 weeks
  Determine the effect of low dose basal insulin detemir (both dependent and independent of weight loss/composition) on relevant metabolic outcomes including:
  insulin sensitivity and beta cell response as measured by oral glucose tolerance test, fasting lipids, markers of inflammation and coagulation, measurements of endothelial function, and neuroendocrine hormones.
  Determine the effect of low dose basal insulin detemir on measures of that are effected by dopamine signaling including depression and mood, cognitive function, feeding related behavior, and personality including impulsivity.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Niswender, MD/PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Lillegard K, Del Castillo JA, Silver HJ. Poorly controlled glycemia and worse beta cell function associate with higher resting and total energy expenditure in adults with obesity and type 2 diabetes: A doubly labeled water study. Clin Nutr. 2024 Mar;43(3):729-738. doi: 10.1016/j.clnu.2024.01.011. Epub 2024 Jan 17. PMID 38320464